CLINICAL TRIAL: NCT00836719
Title: Safety and Neuroprotective Effects of Polyphenon E in Multiple Sclerosis
Brief Title: Safety of Polyphenon E in Multiple Sclerosis Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jesus Lovera MD, Assistant Profesor, Louisiana State University Health Sciences Center in New Orleans
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23AT004433-01 (NIH); K23AT004433-01 (NIH); 1K23AT004433-01 (NIH)
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; safety; open label; Polyphenon E; EGCG; NAA; N-acetyl-aspartate; MRI
MeSH Terms: conditions — Multiple Sclerosis | interventions — polyphenon E; Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Polyphenon E (Experimental): Standarized green tea extract containing 50% EGCG
  Interventions: Drug: Polyphenon E

INTERVENTIONS:
Drug: Polyphenon E — Polyphenon E capsules containing 200 mg of Epigallocachin-galleate. Two capsules twice a day.
  Other Names: EGCG; Green tea extract

SUMMARY:
This study is an open label 6 month study. All subjects will be treated with Polyphenon E (400 mg EGCG twice a day) for six months. The main outcome of this pilot phase will be safety. Secondary outcomes are the change in NAA levels over 6 months as measured by MR-spectroscopy. NAA levels are a marker of neuronal function. We think that Polyphenon E will protect neurons and thus increase NAA levels.

DETAILED DESCRIPTION:
Additional clinical data include changes in EDSS, MS functional composite and cognitive testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS by McDonald criteria
* Relapsing-remitting MS or secondary progressive MS
* Stable therapy with Copaxone, for at least six months prior to inclusion in the study or no therapy for six months in subjects refusing therapy.
* EDSS Score less than or equal to 6.5 (able to walk about 20 meters without resting)
* Ages 18-60.
* Leukocytes ≥3,000/µL
* Absolute neutrophil count ≥1,500/µL
* Platelets ≥100,000/µL
* Total bilirubin ≤local upper limit of normal
* normal AST (SGOT) ALT (SGPT)
* normal serum Creatinine
* women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.
* Willing to drink at most one cup of black tea and two cups of coffee per day, and abstain from drinking green tea or taking supplements containing green tea or green tea compounds, for the duration of the investigation.

Exclusion Criteria:

* MS relapse within the 30 days prior to enrollment.
* A primary progressive form of MS.
* Previous treatment prior to study entry as follows: complete radiation ablation of the bone marrow or anti-CD4 antibody treatment (Campath) at any time; mitoxantrone, cyclophosphamide, cyclosporin, Natalizumab or other immunomodulatory or immunosuppressant therapies except for Copaxone or methylprednisone for relapses within prior nine months.
* History of renal or liver disease.
* Consumption of green tea or supplements containing green tea or tea extract within 30 days prior to enrollment.
* Participants may not participate in any other clinical trial involving investigational agents during the study, or within six months prior to enrolling in the study.
* history of allergic reactions attributed to compounds of similar chemical or biologic composition to Polyphenon E, tea, or any of the inactive ingredients present in the active or placebo capsules, including gelatin.
* history of allergic reactions to gadolinium or any other condition contraindicated for MRI.
* Uncontrolled, clinically-relevant active illness (aside from MS) including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any condition which would make the subject, in the opinion of the investigator, unsuitable for the study.
* Inability to complete the baseline MRI scan.
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus F Lovera, MD, MSPH, Principal Investigator — LSUHSC
Locations (1):
- Louisiana Health Sciences Center New Orleans, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Aktas O, Prozorovski T, Smorodchenko A, Savaskan NE, Lauster R, Kloetzel PM, Infante-Duarte C, Brocke S, Zipp F. Green tea epigallocatechin-3-gallate mediates T cellular NF-kappa B inhibition and exerts neuroprotection in autoimmune encephalomyelitis. J Immunol. 2004 Nov 1;173(9):5794-800. doi: 10.4049/jimmunol.173.9.5794. PMID 15494532
- [Derived] Lovera J, Ramos A, Devier D, Garrison V, Kovner B, Reza T, Koop D, Rooney W, Foundas A, Bourdette D. Polyphenon E, non-futile at neuroprotection in multiple sclerosis but unpredictably hepatotoxic: Phase I single group and phase II randomized placebo-controlled studies. J Neurol Sci. 2015 Nov 15;358(1-2):46-52. doi: 10.1016/j.jns.2015.08.006. Epub 2015 Aug 7. PMID 26298797

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in 9/2009 and ended 4/2010. Subjects were recruited from the LSU MS Clinic and from the community. Advertisements were placed in the quarterly MS Society newsletter and email list.
Groups:
- Polyphenon E: Standarized green tea extract containing 50% EGCG
  Polyphenon E : Polyphenon E capsules containing 200 mg of Epigallocachin-galleate.
  Two capsules twice a day.
Period: Overall Study
Arm/Group | Polyphenon E
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Polyphenon E
Number analyzed (Participants) | 10
Age Continuous [Median (Full Range); unit: years] | 45 [39 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Type of MS [Number; unit: participants]
  Relapsing Remitting | 9
  Secondary Progressive | 1
Expanded Disability Status Scale [Median (Full Range); unit: points] — Expanded Disability Status Scale. Scored according to Neurostatus guidelines.Vakues range from 0-10. Higher values are worse.
  points | 4 [1 to 6.5]
Disease duration [Median (Full Range); unit: years] | 14 [3 to 34]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Serious Adverse Events
Time Frame: six months
Measure: Number; unit: participants
Arm/Group | Polyphenon E
Number analyzed (Participants) | 10
participants | 0

2. Secondary Outcome: Change in Brain NAA Level as Measured by MR Spectroscopy
Description: percent change from baseline to exit in NAA levels adjusted for creatine levels
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percentage change from baseline
Arm/Group | Polyphenon E
Number analyzed (Participants) | 10
percentage change from baseline | 10 [3.4 to 16.2]
Statistical Analysis 1: Comparison: Polyphenon E; N-Acetylaspartate acid (NAA) levels were measured at baseline and exit (6 months). Voxels with less than 30% error in NAA and Creatine (Cre) were used.NAA, Cre and Proton Density were log transformed; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Anisotropic power spatial covariance matrix with terms for time and the registered voxel. Kenward Rogers approx. for degrees of freedom; Mean Difference (Final Values) = 10, 95% CI [3.4 to 16.2] — Dependent variable: NAA. Main effect: visit. Covariates Cre, %GM, %WM, %CSF and %lesion in the voxel

ADVERSE EVENTS:
Arm/Group | Polyphenon E
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyphenon E (N=10)
ALT (Investigations) | 2 (2)
Pain other abdomen NOS (Gastrointestinal disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Skin infection (Infections and infestations) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2)
fatigue (General disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (6)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
restless legs (Nervous system disorders) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
sinusitis (Infections and infestations) | 1 (1)
subconjunctival hemorrage (Eye disorders) | 1 (1)
upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
The study was a pilot study with a small sample size and no control group. The primary endpoint was futility in change in NAA thus the p-values for the primary endpoint are nominal only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No